CLINICAL TRIAL: NCT00004327
Title: Phase II Pilot Study of Octreotide, a Somatostatin Octapeptide Analog, for Gastrointestinal Hemorrhage in Hormone-Refractory Hereditary Hemorrhagic Telangiectasia and Senile Ectasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Yale University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11875; YALESM-7893
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Ectasia
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; hereditary hemorrhagic telangiectasia; rare disease; senile ectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Dilatation, Pathologic; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases | interventions — Octreotide

INTERVENTIONS:
Drug: octreotide

SUMMARY:
OBJECTIVES:

I. Evaluate the efficacy of octreotide, a somatostatin octapeptide analog, in decreasing gastrointestinal bleeding in patients with hormone-refractory hereditary hemorrhagic telangiectasia or senile ectasia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are treated with subcutaneous injections of octreotide twice a day. The dose is adjusted based on response.

If there is no requirement for transfusions or intravenous iron for 4 weeks and the hemoglobin is greater than 10 mg/dL, therapy is continued for 1 year. If there is no decrease in bleeding after 10 weeks, the patient is removed from study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Hereditary hemorrhagic telangiectasia or senile ectasia Refractory to or unable to tolerate hormonal therapy, i.e.: Estrogen Progesterone Danazol Gastrointestinal (GI) hemorrhage requiring transfusion within past 3 months Recurrent GI bleeding over more than 1 year At least 4 units packed RBCs transfused within past year OR intravenous iron required more than 4 times within past year No other likely source of hemorrhage determined within past year --Prior/Concurrent Therapy-- Disease hormone-refractory --Patient Characteristics-- No octreotide sensitivity

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8
Dates: Start 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R. Korzenik, Study Chair — Yale University